CLINICAL TRIAL: NCT04123223
Title: Comparing Cognitive Remediation Approaches for Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Wesleyan University (Other)
Collaborators: Hartford Hospital (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Matthew M. Kurtz, Professor, Wesleyan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R15MH117676-01A1 (NIH); 1R15MH117676-01A1 (NIH)
Record Dates: First submitted 2019-10-03; First posted 2019-10-10 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Cognitive Remediation

STUDY DESIGN:
Intervention Model Description: Cognitive remediation (CR) is a type of behavioral intervention that addresses cognitive deficits in schizophrenia by restoring lost cognitive skills or providing strategies for bypassing deficits through task practice. The present project seeks to identify cognitive training mechanisms that are most effective at improving cognitive function in schizophrenia by comparing two different systematic programs of CR with different foci: drill-and-practice exercises vs. compensatory strategies.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Restorative CR Intervention (Experimental): The restorative remediation intervention will consist of a target of 50 hours (5 hours per week, 1 hour per day, over 3 months) of a sequence of computerized cognitive exercises designed to improve cognitive function through repeated drill-and-practice of exercises largely focused on attention, working memory and verbal episodic memory. Cognitive deficits will be directly targeted by these exercises. Exercises will be started at individually determined levels of difficulty at which each client will be successful, e.g., 80% accuracy. Task difficulty will be increased as performance improves.
  Interventions: Behavioral: Cognitive Remediation
- Strategy CR Intervention (Experimental): Participants in this intervention will be treated for 24 hours (2 hours per week, one day per week over 3 months) with Compensatory Cognitive Training (CCT). The therapy targets four cognitive domains: (a) prospective memory, (b) attention and vigilance, (c) learning and memory, and (d) executive function. The program is a group-based intervention that teaches strategies via interactive, game-like activities to maintain interest and enhance motivation and engagement.
  Interventions: Behavioral: Cognitive Remediation
- Computer Games (Placebo Comparator): Three months of 1-hour, 5-times per week, client-selected computer games.
  Interventions: Behavioral: Computer Games

INTERVENTIONS:
Behavioral: Cognitive Remediation — Cognitive remediation (CR) is a behavioral treatment designed to address neurocognitive deficits through task practice and/or strategy acquisition.
  Arms: Restorative CR Intervention; Strategy CR Intervention
Behavioral: Computer Games — Sham placebo treatment
  Arms: Computer Games

SUMMARY:
This research compares the relative efficacy of two empirically-supported, standardized programs of cognitive remediation for treatment of cognitive deficits and community function in schizophrenia to help inform best practices. The proposed study advances public health by developing and evaluating new behavioral techniques for improving psychosocial outcome in individuals diagnosed with schizophrenia.

DETAILED DESCRIPTION:
Evidence over the past 30 years has revealed that 70-80% of individuals with schizophrenia exhibit marked neurocognitive deficits on measures of attention, learning and memory, problem-solving, language and sensory-motor skill. Particular significance has been attached to these deficits as their severity has been linked to impaired community function, social problem-solving and progress in psychosocial rehabilitation programs. Cognitive remediation (CR) is a type of behavioral intervention that addresses cognitive deficits in schizophrenia by restoring lost cognitive skills or providing strategies for bypassing deficits through task practice. Meta-analyses have revealed that cognitive remediation is a validated approach to improving cognitive function in schizophrenia, however a lack of precision regarding the active elements of the intervention have prevented its recommendation as a standard treatment for the illness. The present three-year proposal seeks to identify cognitive training mechanisms that are most effective at improving cognitive function in schizophrenia by comparing two different systematic programs of CR with different foci: drill-and-practice exercises vs. compensatory strategies. Both programs have strong preliminary empirical support. One-hundred and thirty-five clients diagnosed with schizophrenia or schizoaffective disorder will be randomly assigned to one of three groups: a neuroplasticity-based, drill-and-practice program of computer-assisted cognitive training exercises designed to restore lost cognitive capacity; a manualized strategy training method for bypassing deficits in cognition, or a computer games control condition. Study measures, organized according to an experimental therapeutics approach, with targets distinguished from outcomes, will assess generalization of any observed training effects.

ELIGIBILITY:
Inclusion Criteria:

1. Meeting DSM-5 criteria for schizophrenia or schizoaffective disorder, presenting for intensive outpatient clinical care.
2. Stabilized on atypical antipsychotic medication for a minimum of 2 months prior to entry into the protocol.
3. A minimum of 2 months since discharge from last hospitalization.

   -

Exclusion Criteria:

1. Uncorrected auditory or visual impairment.
2. Mental retardation (Full Scale IQ<70, as estimated by single word-reading from the WRAT and/or evidence of a history of services).
3. Traumatic brain injury with loss of consciousness for more than 10 minutes.
4. Presence or history of any neurologic illness.
5. Lack of proficiency in English
6. Criteria met for concurrent substance dependence,
7. Scoring within 1SD of healthy control performance (from published norms) on measures of visual vigilance, verbal learning, and working memory.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Matrics Consensus Cognitive Battery score (MCCB composite score) | Measures change from study entry, after 3-months of treatment and at a 3-month follow-up.
  The MCCB includes state-of-the-art cognitive probes selected by 74 experts using the RAND panel method. The battery has strong reliability in schizophrenia and includes multiple forms for many subtests to help control for practice effects. Summary T-scores range from 20 to 80 with higher scores indicating better cognitive performance.
UCSD Performance-Based Skills Assessment | Measures change from study entry, after 3-months of treatment and at a 3-month follow-up.
  This standardized performance-based instrument of everyday function, with evidence of reliability and validity in schizophrenia samples, provides information regarding patients' ability to manage information/planning, finance, communications, mobility and household management in role-play situations.Scores range from 0-20 with higher scores indicating better functioning.
Quality of Life Scale | Measures change from study entry, after 3-months of treatment and at a 3-month follow-up.
  A 21-item scale commonly used as a measure of psychosocial functioning in schizophrenia. The Quality-of-Life Scale balances subjective questions regarding life satisfaction and objective indicators of social and occupational role functioning.Scores range from 0-42 with higher scores indicating better functioning.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Institute of Living, Hartford, Connecticut
  - River Valley Services, Middletown, Connecticut